CLINICAL TRIAL: NCT01718405
Title: Genetic Polymorphism as Moderator of the Effect of an Acute Bout of Exercise on Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: 0049
Record Dates: First submitted 2012-10-10; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Executive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise Group (Experimental): Each individual subject will give a blood sample for genetic analysis and undertake an exercise session and a rest session as a control. Cognitive function will be tested before and after each session.
  Interventions: Other: Cognitive function after exercise test; Genetic: Blood sample analysis

INTERVENTIONS:
Other: Cognitive function after exercise test — The individual subjects will participate in 3 sessions of either aerobic exercise, resistance exercise or rest, in a random order. Before and after each session, the subject will take computerized cognitive tests.
Genetic: Blood sample analysis — In the first evaluation session blood samples will be taken from each subject and will be analysed for genetic polymorphism.

SUMMARY:
Studies have shown that an acute bout of aerobic exercise positively effects cognition, mainly executive functioning; however the effect is not observed among all people and it is not clear whether only aerobic exercise can produce this effect or possibly also resistant exercise. The main purpose of our study is to examine whether genetic variation is a moderator of this effect and whether resistant exercise is comparable to aerobic exercise in improving cognition following a single bout of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Physical Education Students
* Able to sign consent form

Exclusion Criteria:

* Competitive athletes
* Smokers
* Neurologic or psychologic orders
* Chronic diseases
* Head Injuries
* Hospitalization in the previous 3 months
* Pregnant

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Cognitive Functioning After Exercise | Five minutes
  Computerized battery of tests evaluating cognitive functioning

OTHER OUTCOMES:
Genetic Variation Associated with Different Cognitive Functioning | Two years
  Genetic variation will be analyzed by extraction of genomic DNA from blood leukocytes, using a salting out procedure, and then by using polymerase chain reaction restriction fragment lengths polymorphism (PCR-RELP) methods for detection of single nucleotide polymorphism. A mutation will be discriminated by digestion with specific restriction endonucleases.

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute, Netanya, Israel